CLINICAL TRIAL: NCT07334951
Title: Effect of AURICULAR Vagus Nerve Stimulation on Glucose Tolerance, and Mood States in Obesity
Brief Title: Effect of Tvns in Obesity
Acronym: TVNS EFFECTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas Wagdy Elsaid Ahmed, Effect of auricular vagus nerve stimulation on glucose tolerance, and mood states in obesity, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TVNS in obesity effects
Record Dates: First submitted 2025-11-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Obesity and Diabetes Mellitus, Type 2
Keywords: Protection from diabetes in obesity
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: They will receive TVNS for 45 min , 3times per week inaddition to dietary advices for months.
Who Masked: Participant
Masking Description: Sham tVNS for 45 min 3 times per week in addition to dietary advices for 3 months .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect of tvns in glucose tolerance ,insulin resistance,stress hormones ,and mood states in obesity (Active Comparator): All patients received transcutaneous electrical nerve stimulation. Allsubsequent ttt will be 3 times per week for 12weeks .
  Patients will also instructed to complete diary booklet each day to describe side effects corresponding with or temporally related to ttt.
  The investigators checked all booklets at the 6 and 12 week assessments. The points for tvns are located in the auricular concha area where there is rich vagus nerve branch distribution.
  Stimulation parameters will be 1MA of electrical current frequency of 20 HZ with pulse duration less than or equal 1ms ,administration once daily lasted 45 min the intensity adjusted based on the individual tolerance of patients.
  Control group Sham tavns ttt location at the superior scapha , where no vagus nerve distribution, after final session, all baseline measurements will be repeated using the same procedures .
  All data will be anonymized and stored securely .data will be verified by double _checked , and analysis by SPSS v26.
  Interventions: Device: Trans vagus nerve stimulation electrical device.
- Control group (Sham Comparator): Sham TVNS 45 min for 3 months with dietary advices .
  Interventions: Device: Trans vagus nerve stimulation electrical device.

INTERVENTIONS:
Device: Trans vagus nerve stimulation electrical device. — Tvns located at auricular concha area For 45min three times per week for 3 months.
  Other Names: TVNS electrical device .

SUMMARY:
Avoid unhealthy foods, walk every day for at least 15 min , sleep well, he should take sessions at its time, family should Avoid disturbances, keep quiet as much as possible, make Analysis recoired before and after interaction.

DETAILED DESCRIPTION:
Pre and post Anthrompometric measurement,waist circumference, body composition, lab tests, mood assessment, tVNS application, data management will be carried out using SPSSv26.

ELIGIBILITY:
Inclusion Criteria:40_50years Both sexes , BMI more than or equal 30 kg/m2 FBG less than 7 mmol/l 2hpp between 7.8 and 11.1mmol/l at the time of enrollment . HOMA-IR >2.9 All are sedentary level activities.

Exclusion Criteria:Diagnostic type 1and 2 DM Cardiovascular disease, stroke, uncontrolled hypertension Use psychoactive drugs, antiepliptic drugs, antidepressants. Present of metal implants, pace maker or cochlear implants. History of epilepsy or seizours . Pregnancy or breast feeding. Dermatologist condition near stimulating site. Major psychiatric disorders.

-

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-11 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance. | Baseline and after 12th weeks of intervention.
  Change in glucose tolerance assessed using 2_hours oral glucose tolerance test (OGTT), expressed as glucose plasma area under curve (AUC), following a75 g oral glucose load.

SECONDARY OUTCOMES:
Insulin resistance. | Baseline and after 12th weeks of intervention.
  Change in insulin resistance assessed using homeostasis model assessment of insulin resistance (HOMA-IR), calculated from fasting plasma glucose tolerance test and fasting insulin levels.
Insulin sensitvity. | Baseline and after 12th weeks of intervention.
  Change in insulin sensitvity assessed using the Matsuda and Defronzo insulin sensitvity index (ISI), derived from oral glucose tolerance values.

OTHER OUTCOMES:
Body mass index | Baseline and after 12 weeks of intervention.
  Change in body mass index calculated as weight in kilograms divided by height in meter square (kg/m2).
Waist circumference. | Baseline and 12 weeks after the intervention.
  Change in waist circumference measured in centimeters at the midpoint between the lowest rib and the ilkac crest
Body fat percentage. | Baseline and after 12 weeks of intervention.
  Change in fat percentage assessed using the sum of four skin fold thickness measurements (tricepes, suprailiac, abdominal ,and thigh) and calculated using sex specific equations.
Stress hormones ( serum cortisol levels ). | Baseline and after 12 weeks of intervention.
  Change in serum cortisol level measured by chemiluminesence immunoassey
Stress hormones ( ACTH ). | Baseline and after 12 weeks of intervention.
  Change in serum ACTH level measured by chemiluminesence immunoassey
Mood states. | Baseline and after 12th weeks of intervention
  Change in mood states assessed using by the profile of mood states _short form (POMS-SF) , using the total mood disturbance score and subscale scores .

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta general hospital, Tanta, Algarbia, Egypt

REFERENCES:
- [Result] Barazzoni R metal 2023 ,aerobic training
- Available data/document: Study Protocol: enaswagdydaib@gmail.com — https://doing.org/10.1016/j.neulet.2021.136393. — No comments